CLINICAL TRIAL: NCT02691273
Title: Applicability of Cellular Application in Diabetes Type 2 Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM01-HMO-CTIL
Record Dates: First submitted 2016-01-20; First posted 2016-02-25 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- breathing technique (Experimental): this arm includes learning breathing technique using the patient's smartphone.
  Interventions: Behavioral: cellular application treating diabetes using breathing technique

INTERVENTIONS:
Behavioral: cellular application treating diabetes using breathing technique

SUMMARY:
It was found that an important part of the factors impeding adherence to medication and a healthy lifestyle among the chronically ill diabetic patients lies in proper management of the disease. Since it is a chronic progressive disease the caregiver is the patient himself.Studies have shown that software system, sending text messages / messages / reminders daily and answering questionnaires can improve adherence to a change in lifestyle.

This study is an initial pilot study , which examines Feasibility ( Applicability ) of using a smart application that promotes a healthy lifestyle perseverance parallel use relaxation techniques .

ELIGIBILITY:
Inclusion Criteria:

* HbA1c above 7.5.
* Smartphone users.
* English and Hebrew literate.

Exclusion Criteria:

*Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
10 percentage improvement in the quality of life questionnaire | two months

CONTACTS AND LOCATIONS:
Overall Officials: Avivit Cohen, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No